CLINICAL TRIAL: NCT07299396
Title: THE EFFECT OF ALVEOLAR RECRUITMENT MANOEUVRE ON INTRAOPERATIVE HAEMODYNAMICS
Status: Completed | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ozlem Sagir, MD, Professor, MD, Balikesir University
Other Study IDs: BalikesirU OSagır 001
Record Dates: First submitted 2025-04-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-04

CONDITIONS: ASA Class I/II Patients Scheduled for Surgery Under General Anesthesia; Laparoscopic Hysterectomy
Keywords: lung protective ventilation; recruitment manoeuvre; laparoscopic surgery; haemodynamic changes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alveolar Recruitment Maneuver Applied
- Alveolar Recruitment Maneuver Not Applied

SUMMARY:
Alveolar recruitment manoeuvre plays a key role in the prevention of atelectasis. In addition, it affects haemodynamic parameters. This study aims to investigate the effects of RM on haemodynamic parameters using minimally invasive monitoring techniques.

DETAILED DESCRIPTION:
During laparoscopic hysterectomy, pneumoperitoneum is created with carbon dioxide (CO₂) to provide surgical field of view and the patient is placed in Trendelenburg position. This increases intrathoracic pressure, decreases lung compliance and increases the risk of atelectasis. Therefore, lung protective ventilation strategies such as alveolar recruitment manoeuvre (RM), individualised PEEP application and low tidal volume are recommended. RM aims to increase lung compliance and prevent atelectasis by reopening collapsed alveoli. However, changes in haemodynamic parameters, especially mean arterial pressure and cardiac output, may occur during RM. In addition to standard monitoring for the management of these changes, haemodynamic evaluation can be performed with minimally invasive methods such as arterial waveform analysis. In this study, we aimed to evaluate the effects of RM applied during laparoscopic hysterectomy on intraoperative haemodynamic parameters using arterial waveform analysis.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class 1-2 patients 18-70 years old

Exclusion Criteria:

* <18 y, BMI>40
* Patients receiving invasive mechanical ventilator support in the last 1 month
* Patients who have received chemotherapy or radiotherapy in the last 2 months
* Those with severe lung disease (COPD, asthma, pulmonary infection, bronchiectasis, previous need for non-invasive mechanical ventilation, oxygen therapy or steroid therapy for acute attack)
* Known severe pulmonary hypertension
* Patient refusal to participate in the study
* Intracranial tumour
* Haemodynamic instability
* Shock
* Neuromuscular disease
* Pathologies causing increased intracranial and intraocular pressure
* Atrial fibrillation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — laparoscopic hysterectomy patients
Study Population: * ASA I-II risk group patients
  * Patients between 18-70 y undergoing laparoscopic hysterectomy surgery
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Effect of RM on heart rate (in bpm) | perioperatively
  measurement of heart rate in bpm
Effect of RM on pressure mmHg | perioperatively
  blood pressure measurement in mmmercury
Effect of RM on Cardiac index(CI) | intraoperatively
  Cardiac Index measurement via an arterial cannula as l/min/m2
Effect of RM on stroke volume index(SVI) | intraoperatively
  SVI measurement via arterial cannula as L/min/m2
Effect of RM on pulse pressure variablity(PPV) | intraoperatively
  pulse pressure variability measured by finger probe as cm/s
Effect of RM on systemic vascular resistance index(SVRI) | intraoperatively
  systemic vascular resistance index(SVRI) measurement via arterial cannula as L/min/m2
Effect of RM on cardiac power index(CPI) | intraoperatively
  cardiac power index(CPI) measurement via arterial line as ml/min/m2

SECONDARY OUTCOMES:
Effect of RM on Compliance | intraoperatively
  measurement of dynamic compliance by Ventilator as Cdyn
Effect of RM on Oxygenation | İntraoperatively
  measurement of oxygenation via obtaining partial blood oxygene pressure via arterial blood sample pulse oxymeter as %
Postoperative pulmonary comlications (infection, bronchospasm, pleural effusion, atelectasis, respiratory failure) | postoperative day 1 and 3
  assessment of pulmonary complications

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Koroglu, Professor, medical doctor, Study Chair — Balikesir University
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes